CLINICAL TRIAL: NCT02957149
Title: A Study Evaluating Intraoperative Application of Platelet-Rich Plasma to the Neurovascular Bundles During Nerve-Sparing Radical Prostatectomy: Initial Technical Description and Prospective Early Postoperative Outcomes Analysis
Brief Title: Platelet Rich Plasma During Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC2051; MC2051 (Other: Mayo Clinic); NCI-2020-00836 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-001320 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Platelet Rich Plasma (PRP) Treatment (Experimental): Platelets that are collected from the subject during the radical prostatectomy, for prostate cancer. The Autologous Platelet-Rich Plasma is concentrated in a device (Angel Concentrated Platelet Rich Plasma System) to 1,000,000 platelets/mL and applied topically once to the neurovascular bundle during the surgery.
  Interventions: Other: Autologous Platelet-Rich Plasma; Device: Angel Concentrated Platelet Rich Plasma System

INTERVENTIONS:
Other: Autologous Platelet-Rich Plasma — Platelets that are collected from the subject during the radical prostatectomy, for prostate cancer. The platelets are concentrated in a device to 1,000,000 platelets/mL and applied topically once to the neurovascular bundle during the surgery.
  Other Names: PRP
Device: Angel Concentrated Platelet Rich Plasma System

SUMMARY:
Can platelet rich plasma applied to nerve bundles at time of surgery help the nerve bundles heal? Subjects undergoing a Radical Prostatectomy who meet study inclusion/exclusion criteria will be consented to receive an intraoperative application of platelet-rich plasma, made from their own blood at the time of surgery, for application onto their neurovascular bundles in an effort to improve the healing process. Subjects will be followed for an additional 18 months to determine the efficacy and safety of this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, clinically localized prostatic adenocarcinoma
* Age 50 - 60 years
* Male gender
* Normal preoperative sexual function
* Normal urinary continence

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Vulnerable study populations
* Active systemic infection
* Diabetes mellitus diagnosis
* Preexisting Erectile Dysfunction or urinary incontinence
* Metastatic or locally advanced prostatic adenocarcinoma on preoperative evaluation
* Men found grossly or pathologically to have locally advanced or metastatic disease at the time of radical prostatectomy
* An estimated blood loss of > 750 mL at the time of radical prostatectomy
* Treatment prior to surgery with any form of hormones, anti-androgens or androgen deprivation therapy
* Use of an antidepressant, beta blocker or erectile dysfunction medication at the time of study screening
* Men without a regular sexual partner
* Use of aspirin or heparin 2 weeks before radical prostatectomy
* Need for use of aspirin or heparin for 2 weeks or more after radical prostatectomy

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T. Gettman, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Platelet Rich Plasma (PRP) Treatment: Platelets that are collected from the subject during the radical prostatectomy, for prostate cancer. The Autologous Platelet-Rich Plasma is concentrated in a device (Angel Concentrated Platelet Rich Plasma System) to 1,000,000 platelets/mL and applied topically once to the neurovascular bundle during the surgery.
  Autologous Platelet-Rich Plasma: Platelets that are collected from the subject during the radical prostatectomy, for prostate cancer. The platelets are concentrated in a device to 1,000,000 platelets/mL and applied topically once to the neurovascular bundle during the surgery.
  Angel Concentrated Platelet Rich Plasma System
Period: Overall Study
Arm/Group | Platelet Rich Plasma (PRP) Treatment
Started | 24
Completed | 19
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Platelet Rich Plasma (PRP) Treatment
Number analyzed (Participants) | 19
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [57 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Safety of Using Platelet Rich Plasma (PRP) on the Neurovascular Bundle (NVB)
Description: Assessed by the number of subjects experiencing serious adverse events (SAEs) after treatment with PRP following nerve-sparing radical prostatectomy
Time Frame: 18 months
Population: The highest grade of adverse event (AE) is reported for each participants who experienced one or more AE.
Measure: Count of Participants; unit: Participants
Arm/Group | Platelet Rich Plasma (PRP) Treatment
Number analyzed (Participants) | 19
Participants
  Grade 3 or higher AE (severe or life-threatening) | 0
  Grade 1 or 2 AE (mild or moderate) | 2
  No AE | 17

2. Secondary Outcome: Change in Sexual Function Using International Index of Erectile Function (IIEF-5)
Description: The IIEF-5 (International Index of Erectile Function) is used for diagnosis of erectile dysfunction (ED). The IIEF-5, also knows as the Sexual Health Inventory for Men (SHIM), is a 5-question survey designed to assess the presence and severity of ED over the past 6 months. Questions are answered on a scale of 1-5. A score of 21 or lower is often considered indicative of ED. The IIEF-5 classifies ED into five categories based on scores: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25).
Time Frame: Baseline; every 3 months up to 18 months.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Platelet Rich Plasma (PRP) Treatment
Number analyzed (Participants) | 19
score on a scale
  Baseline | 25 [25 to 25]
  3 months | 16 [8.5 to 20]
  6 months | 19 [12.5 to 21.5]
  9 months | 19 [14 to 21.5]
  12 months | 20 [18 to 24]
  18 months | 20 [18 to 22.5]

3. Secondary Outcome: Change in Urinary Function (UF) Using the Expanded Prostate Cancer Index Composite (EPIC)
Description: The Urinary Function (UF) section of the Expanded Prostate Cancer Index composite (EPIC) questionnaire consists of 7 questions evaluating urinary habits over the past 4 weeks. To assess change in UF over time, evaluation focused on response to question 5 (number of pads or adult diapers used to control leakage), with normal urinary continence defined as a response of "none" per protocol. Responses are recorded on a scale of 0-3 where 0=None, 1=1 pad per day; 2=2 pads per day; and 3=3 or more pads per day.
Time Frame: Baseline; 3 months; 6 months; 9 months; 12 months; 18 months
Population: 4 patients were lost to follow-up for the last visit (18 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Platelet Rich Plasma (PRP) Treatment
Number analyzed (Participants) | 19
Participants
  Baseline | 18
  3 Months | 9
  6 Months | 15
  9 Months | 18
  12 Months | 18
  18 Months: number analyzed (Participants) | 15
  18 Months | 15

ADVERSE EVENTS:
Time Frame: 18 months
Description: Patients were followed from enrollment up to 18 months. We grade all the AEs using the CTCAE. 2 patients developed an AE, one patient experienced 2 grade 1 AEs and a single grade 2 AE; the second patient had a single grade 2 AE.
Arm/Group | Platelet Rich Plasma (PRP) Treatment
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 2/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platelet Rich Plasma (PRP) Treatment (N=19)
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Grade 1
Interstitial Cystitis (Acute) (Renal and urinary disorders) | 1 (1) — Grade 1
Hematuria (Renal and urinary disorders) | 1 (1) — Grade 2
Dysuria (Renal and urinary disorders) | 1 (1) — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT02957149/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT02957149/ICF_001.pdf